CLINICAL TRIAL: NCT04224701
Title: A Randomized, Double-blinded, Placebo-controlled, Dose-escalation Phase 1 Clinical Trial to Evaluate the Safety and Immunogenicity of Recombinant HIV-1 Envelope Protein BG505 SOSIP.GT1.1 Gp140 Vaccine, Adjuvanted in Healthy, HIV-uninfected Adults
Brief Title: A Clinical Trial to Evaluate the Safety and Immunogenicity of Recombinant HIV-1 Envelope Protein BG505 SOSIP.GT1.1 Gp140 Vaccine, Adjuvanted in Healthy, HIV-uninfected Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: International AIDS Vaccine Initiative (Network)
Collaborators: GlaxoSmithKline (Industry); Rockefeller University (Other); George Washington University (Other); Amsterdam UMC, location VUmc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: IAVI C101
Record Dates: First submitted 2019-12-19; First posted 2020-01-13 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Investigational Product, 30 µg/ Placebo (Experimental): 30 µg IM, months 0, 2 and 6
  Interventions: Biological: BG505 SOSIP GT1.1 gp140 Vaccine, Adjuvanted; Biological: Placebo
- Investigational Product, 300 µg/ Placebo (Experimental): 300 µg IM, months 0, 2 and 6
  Interventions: Biological: BG505 SOSIP GT1.1 gp140 Vaccine, Adjuvanted; Biological: Placebo

INTERVENTIONS:
Biological: BG505 SOSIP GT1.1 gp140 Vaccine, Adjuvanted — 30 µg
  Arms: Investigational Product, 30 µg/ Placebo
Biological: BG505 SOSIP GT1.1 gp140 Vaccine, Adjuvanted — 300 µg
  Arms: Investigational Product, 300 µg/ Placebo
Biological: Placebo — Tris NaCl Diluent

SUMMARY:
This is a phase 1 clinical trial to evaluate the safety, tolerability, and immunogenicity of HIV-1 envelope protein BG505 SOSIP.GT1.1 gp140 trimer Vaccine, Adjuvanted, in up to 48 healthy HIV-uninfected adult volunteers.

DETAILED DESCRIPTION:
This is a phase 1 clinical trial to evaluate the safety, tolerability, and immunogenicity of HIV-1 envelope protein BG505 SOSIP.GT1.1 gp140 trimer Vaccine, Adjuvanted, in up to 48 healthy HIV-uninfected adult volunteers. BG505 SOSIP.GT1.1 is a soluable, cleavage-competent, trimeric HIV-1 envelope glycoprotein gp140 formulated in 0.55mL at 2mg/mL in 20 mM Tris, 100 mM naCL, pH 7.5 and will be administered IM.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults as assessed by a medical history, physical exam, and laboratory tests;
2. At least 18 years of age on the day of screening and has not reached his/her 51 birthday on the day of first IP administration;
3. Willing to comply with the requirements of the protocol and be available for follow-up for the planned duration of the study;
4. In the opinion of the Principal Investigator or designee and based on Assessment of Informed Consent Understanding results, has understood the information provided and potential impact and/or risks linked to IP administration and participation in the trial; written informed consent will be obtained from the volunteer before any study-related procedures are performed;
5. Willing to undergo HIV testing, risk reduction counseling and receive HIV test results;
6. All volunteers born female who are engaging in sexual activity that could lead to pregnancy must commit to use an effective method of contraception at the time of the first IP administration and for 4 months following the last IP administration.
7. All volunteers born female who are not heterosexually active at screening must agree to utilize an effective method of contraception if they become heterosexually active as outlined above;
8. All volunteers born female must be willing to undergo urine pregnancy tests at time points indicated in the Schedule of Procedures
9. All sexually active volunteers born male, regardless of reproductive potential, must be willing to use an effective method of contraception (such as consistent condom use) from the day of the first IP administration until at least 4 months after the last IP administration;
10. Willing to forgo donations of blood, or any other tissues during the study and, for those who test HIV-positive due to IP-induced antibodies, until the anti-HIV antibody titers become undetectable.
11. For sites in the European Union (EU), consent to the collection and use of personal data in compliance with the General Data Protection Regulation (GDPR)

Exclusion Criteria:

1. Confirmed HIV-1 or HIV-2 infection;
2. Any clinically relevant abnormality on history or examination, including history of immunodeficiency or autoimmune disease; use of systemic corticosteroids (the use of topical or inhaled steroids is permitted), immunosuppressive, anticancer, antituberculosis or other medications considered significant by the investigator within the previous 6 months;
3. Any clinically significant acute or chronic medical condition that is considered progressive or in the opinion of the investigator makes the volunteer unsuitable for participation in the study;
4. Reported behavior which put the volunteer at risk for HIV infection within 6 months prior to IP administration, as defined by:

   * Unprotected sexual intercourse with a known HIV-infected person, a partner known to be at high risk for HIV infection or a casual partner (i.e., no continuing established relationship)
   * Engaged in sex work
   * Frequent excessive daily alcohol use or frequent binge drinking, or any other use of illicit drugs
   * History of newly-acquired syphilis, gonorrhea, non-gonococcal urethritis, HSV-2, chlamydia, pelvic inflammatory disease (PID), trichomonas, mucopurulent cervicitis, epididymitis, proctitis, lymphogranuloma venereum, chancroid, or hepatitis B or hepatitis C;
   * Three or more sexual partners
5. If female, pregnant or planning a pregnancy during the period of enrolment until 4 months after the last IP administration; or lactating;
6. Bleeding disorder that was diagnosed by a physician (e.g., factor deficiency, coagulopathy or platelet disorder that requires special precautions)
7. Infectious disease diagnosis: chronic hepatitis B infection (HbsAg-positive), current hepatitis C infection (HCV Ab positive and HCV RNA positive or interferon-alfa treatment for hepatitis C infection in the past year or interferon-alfa-free treatment for hepatitis C infection completed in the past 6 months), or active syphilis (screening and confirmatory tests);
8. History of splenectomy;
9. Any of the following abnormal laboratory parameters listed below:

   Hematology
   * Hemoglobin - <10.5 g/dl or <6.5 mmol/L in females; <11.0 g/dl or <6.8 mmol/L in males
   * Absolute Neutrophil Count (ANC) - ≤1,000/mm3 or < 1.0 x 109 cells/L
   * Absolute Lymphocyte Count (ALC) - ≤650/mm3 or < 0.65 x 109 cells/L
   * Platelets - <125,000 cells/mm3 or < 125 x 109 cells/L

   Chemistry
   * Creatinine - >1.1 x upper limit of normal (ULN)
   * AST - >1.25 x ULN
   * ALT - >1.25 x ULN

   Urinalysis

   Clinically significant abnormal dipstick confirmed by microscopy:
   * Protein = 1+ or more
   * Blood = 2+ or more (not due to menses)
10. Receipt of live attenuated vaccine within the previous 30 days or planned receipt within 30 days after IP administration; or receipt of other vaccine within the previous 14 days or planned receipt within 14 days after IP administration. (Exception is live attenuated influenza vaccine within 14 days.);
11. Receipt of blood transfusion or blood-derived products within the previous 3 months;
12. Participation in another clinical trial of an investigational product currently, within the previous 3 months or expected participation during this study; concurrent participation in an observational trial not requiring blood or tissue sample collection is not an exclusion;
13. Prior receipt of any investigational HIV vaccine candidate or HIV monoclonal antibody Note: receipt of placebo in a previous HIV vaccine trial or monoclonal antibody trial will not exclude a volunteer from participation if documentation is available and the Medical Monitor gives approval;
14. History of significant local or systemic reactogenicity to vaccines (e.g., anaphylaxis, respiratory difficulties, angioedema, injection site necrosis or ulceration);
15. Psychiatric condition that compromises safety of the volunteer and precludes compliance with the protocol. Specifically excluded are persons with psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years;
16. Seizure disorder: A volunteer who has had a seizure in the last 3 years is excluded. (Not excluded: a volunteer with a history of seizures who has neither required medications nor had a seizure for 3 years);
17. History of malignancy in the past 5 years (prior to screening) or ongoing malignancy (a history of completely excised malignancy that is considered cured is not an exclusion);
18. Active, serious infections requiring antibiotic, antiviral or antifungal therapy within 30 days prior to enrolment;
19. Body mass index (BMI) ≥35;
20. Body weight <110 pounds (50 kg);
21. Prior daily use of NSAID/aspirin that cannot be held for 5 days prior to the leukapheresis procedure (if required by the study site);
22. If, in the opinion of the Principal Investigator, it is not in the best interest of the volunteer to participate in the trial.

Ages: 18 Years to 51 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2023-08-02 (Actual)

PRIMARY OUTCOMES:
Safety - reactogenicity | 7 Days
  Proportion of volunteers with Grade 2 or greater reactogenicity (i.e., solicited adverse events) from Day 0 through Day 7 after each investigational product (IP) administration
Safety - IP related unsolicited adverse events | 28 days
  Proportion of volunteers with IP-related unsolicited adverse events (AEs), including safety laboratory (biochemical, hematological) parameters, from the day of each IP administration up to 28 days post each IP administration
Safety - Grade 2 or greater unsolicited AEs | 28 days
  Proportion of volunteers with Grade 2 or greater unsolicited adverse events (AEs), including safety laboratory (biochemical, hematological) parameters, from the day of each IP administration up to 28 days post each IP administration
Safety - IP related SAEs | 18 Months
  Proportion of volunteers with IP-related serious adverse events (SAEs) throughout the study period
Safety - pIMDs | 18 Months
  Proportion of volunteers in each group with potential immune-mediated diseases (pIMDs) from the day of first IP administration throughout the study period

SECONDARY OUTCOMES:
Immunogenicity - Frequency Ab responses | 6 Months
  Frequency of binding antibody responses to GT1.1 trimer after the first, second, and/or third IP administrations compared to baseline
Immunogenicity - Magnitude Ab responses | 6 Months
  Magnitude of binding antibody responses to GT1.1 trimer after the first, second, and/or third IP administrations compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Marina Caskey, MD, Principal Investigator — Rockefeller University; Godelieve de Bree, MD, PhD, Principal Investigator — Amsterdam UMC, location VUmc; David Joseph Diemert, MD, Principal Investigator — George Washington University
Locations (3):
- United States (2):
  - George Washington University, Washington D.C., District of Columbia
  - Rockefeller University, New York, New York
- The Amsterdam University Medical Centers, Amsterdam, Netherlands

REFERENCES:
- [Derived] Libera M, Caputo V, Laterza G, Moudoud L, Soggiu A, Bonizzi L, Diotti RA. The Question of HIV Vaccine: Why Is a Solution Not Yet Available? J Immunol Res. 2024 Apr 8;2024:2147912. doi: 10.1155/2024/2147912. eCollection 2024. PMID 38628675
- See also: Related Info — http://iavi.org